CLINICAL TRIAL: NCT01118065
Title: A Phase II Study to Investigate the Efficacy of RAD001 (Afinitor®, Everolimus) in Patients With Irresectable Recurrent or Metastatic Differentiated, Undifferentiated (Anaplastic) and Medullary Thyroid Carcinoma
Brief Title: Everolimus in Treating Patients With Progressive or Recurrent, Unresectable, or Metastatic Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: DUT-LUMC-CRAD001CNL08T; CDR0000672171 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2009-016669-27; EU-21037; NL-31245-058-10
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2010-05

CONDITIONS: Head and Neck Cancer
Keywords: anaplastic thyroid cancer; recurrent thyroid cancer; stage III follicular thyroid cancer; stage III papillary thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer; thyroid gland medullary carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — Everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well everolimus works in treating patients with progressive or recurrent, unresectable, or metastatic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of everolimus in patients with progressive or recurrent, unresectable, or metastatic differentiated thyroid carcinoma.

Secondary

* To determine maximum percentage of tumor reduction in these patients.
* To describe activity time to event endpoints.
* To assess toxicity.
* To determine evolution of serum thyroglobulin.
* To perform explorative pharmacogenomic, pharmacokinetic, and translational studies. (exploratory)
* To investigate efficacy of everolimus in patients with progressive or recurrent, unresectable or metastatic disease of undifferentiated (anaplastic) or medullary thyroid cancer.

OUTLINE: Patients receive oral everolimus once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of thyroid cancer meeting ≥ 1 of the following criteria:

  * Progressive or recurrent disease
  * Metastatic disease
  * Unresectable disease
* Meeting any of the following thyroid cancer subtypes:

  * Differentiated thyroid cancer (i.e., papillary, follicular, or Hurthle cell disease) that is radio-iodine refractory
  * Undifferentiated thyroid cancer (i.e., anaplastic disease)
  * Medullary thyroid cancer
* Must have received prior everolimus or other mTOR inhibitor therapy
* Patients with history of brain metastasis who are neurologically stable following definitive radiation and/or surgery and do not require corticosteroids allowed

PATIENT CHARACTERISTICS:

* Karnofsky performance score 70-100%
* ANC ≥ 1,500/mm^³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 5.6 mmol/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for known liver metastases)
* Serum creatinine ≤ 2 times ULN
* Negative pregnancy test
* No other malignancy, except nonmelanoma skin cancer, carcinoma in situ of the cervix, or a malignancy diagnosed and with no current evidence of malignancy within the past 2 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Maximum percentage of tumor reduction
Activity time to event endpoints
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kapiteijn, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] de Wit D, Schneider TC, Moes DJ, Roozen CF, den Hartigh J, Gelderblom H, Guchelaar HJ, van der Hoeven JJ, Links TP, Kapiteijn E, van Erp NP. Everolimus pharmacokinetics and its exposure-toxicity relationship in patients with thyroid cancer. Cancer Chemother Pharmacol. 2016 Jul;78(1):63-71. doi: 10.1007/s00280-016-3050-6. Epub 2016 May 11. PMID 27169792